CLINICAL TRIAL: NCT06641674
Title: Development and Clinical Translation of EGFR Mutation Targeting PET Probe
Brief Title: EGFR Mutation Targeting Molecular Probe for PET Imaging
Acronym: EGFR-PET
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2024YJZ02
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Cancer
Keywords: PET imaging; EGFR mutation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: 18F-LF13 — 18F-LF13 PET/CT: after intravenous injection of 1.85 - 3.7 MBq/kg body weight of quality-controlled 18F-LF13, a Siemens Biograph PET/CT scan will be applied within 0.5 h, and the scan range will be from the top of the head to 1/3 of the upper thigh, 2 h to 4 h delayed scanning can be added if necessary.

SUMMARY:
In this project, investigators plan to develop a F-18 labeled molecular probe in order to detect the EGFR mutation tumor lessions in patients to identify patients benefiting fromTKIs treatment, and evaluate its efficacy in detecting EGFR Del 19 mutant lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female, aged 18-75 years old (including 18 and 75 years old), ECOG score 0 or 1.
2. Patients could understand and sign the informed consent form voluntarily with good compliance.
3. Patients with histologically or cytologically or clinically confirmed lung cancer with measurable disease.
4. Women had to be using an effective contraceptive method (effective contraceptive means sterilisation, intrauterine hormonal devices, condoms, contraceptives/pills, sexual abstinence, or partner's removal of the vas deferens) during the study and for 6 months after the study. Men should consent to subjects who must use contraception during the study period and for 6 months after the end of the study period.
5. Predicted survival greater than 3 months;

Exclusion Criteria:

1. Severe hepatic or renal dysfunction;
2. Pregnant or nursing;
3. Known allergy to the investigational drug or its excipients in study;
4. Unable to comply with the PET/CT imaging procedures;
5. Claustrophobia or other psychiatric disorders;
6. Other conditions deemed unsuitable for participation in the trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lung cancer patients or lung cancer patients treated with TKIs
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard Uptake Value Value | 1 year
  The standardized uptake value (SUV) of 18F-LF13 in EGFR mutation lesion measured by PET/CT

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No